CLINICAL TRIAL: NCT02241512
Title: IV Ibuprofen for the Prevention of Post-ERCP Pancreatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David M Troendle, Dr., University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU 082014-033
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: post-ERCP pancreatitis; pediatric; ibuprofen
MeSH Terms: interventions — Ibuprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental): Single dose IV Ibuprofen at a dose of 10mg/kg (max: 800mg).
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Single dose IV normal saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ibuprofen
  Other Names: Caldolor
  Arms: Ibuprofen
Drug: placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an advanced endoscopic technique utilized to diagnose and treat pathologic conditions involving the ducts draining the liver and pancreas. Post-ERCP pancreatitis (PEP) is the most common complication following ERCP and occurs in approximately 11% of children undergoing the procedure. By definition it leads to prolongation of hospital stay or delays in care and rarely can result in long-term morbidity or even death. Recent adult trials have demonstrated prevention of PEP with administration of rectal nonsteroidal anti-inflammatory drugs (NSAIDS). To date, no studies have been performed in children thus no "gold standard" or even commonly accepted method of preventing PEP in the pediatric population exist. Studying an IV NSAID such as ibuprofen has distinct advantages over rectally administered NSAIDs in the pediatric population in that it would allow for more consistent weight based dosing and would have more predictable absorption compared to suppository. Thus, this project proposes a pilot study evaluating the effectiveness of IV ibuprofen at preventing PEP in the pediatric population. The design of the proposed study is a prospective randomized double-blind trial comparing IV Ibuprofen to placebo controls (normal saline) at the time of procedure in patients undergoing ERCP at Children's Medical Center Dallas over a two-year period. The primary outcome measurement will be development of PEP. Post-ERCP bleeding and change in pre- and post- procedural pain scores will also be measured. The hypothesis is that IV Ibuprofen administered at the time of ERCP will decrease rates of post-ERCP pancreatitis in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age<=18 years
* Undergoing ERCP (defined as cannulation of the major or minor papilla) for any indication

Exclusion Criteria:

* Age>18
* Pancreatitis within the 72 hours preceding ERCP
* Allergy or hypersensitivity to Aspirin or NSAID medications
* Pregnancy or breastfeeding mother
* Cr >1.4
* Gastrointestinal hemorrhage in preceding 72 hours
* Heart disease reliant upon a patient ductus arteriosis
* History of sickle cell disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Troendle, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center of Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Troendle DM, Gurram B, Huang R, Barth BA. IV Ibuprofen for Prevention of Post-ERCP Pancreatitis in Children: A Randomized Placebo-controlled Feasibility Study. J Pediatr Gastroenterol Nutr. 2020 Jan;70(1):121-126. doi: 10.1097/MPG.0000000000002524. PMID 31651801

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients excluded after enrollment. 5 did not undergo ERCP and thus did not receive a study drug. 3 did not have study drug available in time for procedure. 2 did not meet inclusion criteria.
Groups:
- Ibuprofen: Single dose IV Ibuprofen at a dose of 10mg/kg (max: 800mg).
  Ibuprofen
- Placebo: Single dose IV normal saline
  placebo
Period: Overall Study
Arm/Group | Ibuprofen | Placebo
Started | 30 | 29
Completed | 29 | 29
Not Completed | 1 | 0
Not completed — Pump malfunction, drug not delivered | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 29 | 58
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Mean Pain Score [Mean (Inter-Quartile Range); unit: units on a Likert scale] — Baseline pain score on 10-point Likert scale
  units on a Likert scale | 2.9 [0 to 4.5] | 2.2 [0 to 4.0] | 2.6 [0 to 4.5]

OUTCOME MEASURES:

1. Primary Outcome: Post-ERCP Pancreatitis
Description: Number of patients who develop post-ERCP pancreatitis
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 2 | 5

2. Secondary Outcome: Post-ERCP Bleeding
Description: Number of patients who develop post-ERCP bleeding
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 2 | 0

3. Other Pre Specified Outcome: Increased Pain Score
Description: Number of patients with increased pain scores after the procedure
Time Frame: pre-procedural, 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 29 | 29
Participants | 1 | 11

4. Other Pre Specified Outcome: 24-h Post-ERCP Pain Score
Description: Pain score recorded 24-hrs after the ERCP was performed as recorded on a 10-point Likert pain scale (0= lowest value, no pain, 10=highest value, severe pain)
Time Frame: pre-procedural, 24 hours
Measure: Mean (Inter-Quartile Range); unit: score on a Likert pain scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 29 | 29
score on a Likert pain scale | 1.1 [0 to 2] | 3.1 [0 to 6.0]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: All adverse events were defined by the American Society of Gastroenterology (ASGE) lexicon for endoscopic adverse events.
Arm/Group | Ibuprofen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 3/29 | 9/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibuprofen (N=29) | Placebo (N=29)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 5 (5) — Post-ERCP Pancreatitis
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) — Abdominal pain not related to post-ERCP pancreatitis
Bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0) — post-ERCP bleeding
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Post-ERCP cholangitis
Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) — ERCP related perforation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT02241512/Prot_SAP_000.pdf